CLINICAL TRIAL: NCT00517686
Title: Feedback of Treatment Intensification Data to Reduce Cardiovascular Disease Risk (FIT)
Acronym: FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: RFA-HS-07-002
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Cardiovascular Disease (CVD) Risk Factors
Keywords: Poor risk factor control; Treatment intensification; Medication adherence; Cardiovascular disease (CVD)
MeSH Terms: conditions — Cardiovascular Diseases; Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The study will use automated databases and PHASE information systems to identify patients and incorporate feedback on a monthly basis into the ongoing reports used by program staff at facilities randomized to this intervention arm (n=4).
  Interventions: Other: Information feedback intervention
- 2 (No Intervention): Usual care facilities (n=4) will continue to use current PHASE reports that include information on recent risk factor levels and current use of selected medications but no treatment intensification information, and no information on medication adherence.

INTERVENTIONS:
Other: Information feedback intervention — This study will evaluate an information feedback intervention: measuring, reporting and feeding back information to primary care teams on the need for treatment intensification in patients at high risk for cardiovascular disease (CVD).
  Arms: 1

SUMMARY:
The primary research question of this study is to determine whether measuring, reporting and feeding back information to primary care teams on the need for treatment intensification in patients at high risk for cardiovascular disease (CVD) can improve rates of treatment intensification and reduce levels of poorly controlled systolic blood pressure, LDL-c, and A1c.

DETAILED DESCRIPTION:
Project Description: We propose a cluster randomized trial intervention involving eight or more medical facilities of Kaiser Permanente Northern California (KP) and more than 65,000 patients at high risk for CVD. At intervention facilities, patient-level information obtained from KP's electronic health record on the need for treatment intensification (for systolic blood pressure, LDL-c, and A1c) and on recent medication adherence are added to a population management database and fed back through software currently used by staff working with primary care providers. Staff at control facilities continue to use the same population management database and software but only receive information on risk factor levels and selected medications.

Specific Aims:

1. Evaluate the effectiveness of measurement and feedback of treatment intensification information in patients at high risk of CVD for improving rates of treatment intensification and for reducing levels of poorly controlled systolic blood pressure, LDL-c, and A1c.
2. Evaluate the impact of the intervention, compared with current practice, on total numbers of patient contacts, outpatient visits, and costs of care in relation to improvements in risk factor control.
3. Evaluate the effect of this innovation on physician and staff perceptions of the value (effectiveness and efficiency) of the population management program for high-risk patients.

Relevance: If this translational study shows that feedback of information on treatment intensification leads to higher rates of intensification and improved risk factor control, this finding will have shown a population-level use of health information technology for improving clinical quality and will also have validated treatment intensification as a metric of clinical quality.

ELIGIBILITY:
Inclusion Criteria:

Among the randomized medical facilities, we will study a population that is drawn from the PHASE registry and includes patients with at least one of the following:

* Diabetes, coronary artery disease; congestive heart failure; stroke/tia; peripheral artery disease; chronic kidney disease; hypertension; or hyperlipidemia
* PHASE patients must be in poor control for at least one CVD risk factor and meet study criteria for needing treatment intensification at some point during the 6-month period.

Exclusion Criteria:

* All patients eligible for the study will be included in the analyses
* There will be no exclusions based on clinical or other criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16584 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Tightly-linked processes (i.e., was treatment intensified more frequently) measured in the 3 months after initial reporting of need for intensification; and mean levels of intermediate outcomes (SBP, LDL-c, and A1c), measured for all study population. | 3 months; 1 year

SECONDARY OUTCOMES:
Proportions in control for each risk factor; treatment intensification and risk factor improvements in subgroups; and efficiency in terms of patient contacts, visits and costs per unit improvement in risk factor control. | 3 months; 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joe V Selby, MD, MPH, Principal Investigator — Kaiser Permenante, Division of Research
Locations (1):
- Kaiser Permanente - Division of Research, Oakland, California, United States

REFERENCES:
- [Derived] Selby JV, Schmittdiel JA, Fireman B, Jaffe M, Ransom LJ, Dyer W, Uratsu CS, Reed ME, Kerr EA, Hsu J. Improving treatment intensification to reduce cardiovascular disease risk: a cluster randomized trial. BMC Health Serv Res. 2012 Jul 2;12:183. doi: 10.1186/1472-6963-12-183. PMID 22747998